CLINICAL TRIAL: NCT03598101
Title: TONEFITreha: Proof of Concept and Usability of a Portable Exercise Device to Improve Cardiovascular Functioning and Balance in Neuro-orthopaedic Rehabilitation.
Brief Title: TONEFITreha: Proof of Concept and Usability Study.
Acronym: TONFITreha
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reha Rheinfelden (Other)
Responsible Party: Principal Investigator, Frank Behrendt, Principal Investigator, Reha Rheinfelden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-00793
Record Dates: First submitted 2018-06-18; First posted 2018-07-26 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Neurological Disorder; Orthopedic Disorder
MeSH Terms: conditions — Nervous System Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental)
  Interventions: Device: TONEFITreha

INTERVENTIONS:
Device: TONEFITreha — The newly developed Tonefit Reha is based on the existing fitness device, the TONEFIT belt. Similar to Nordic Walking, the device aims to include upper limb activity in walking exercise to train the shoulder girdle and arm. While Nordic Walking uses poles, the existing TONEFIT belt uses body-worn resistance handles to actively involve the upper body. It is worn around the waist, like a belt. The two independent pull-push elements with non-adjustable resistance on each side allow increased intensity for strengthening and endurance training during walking, particular for upper extremities and trunk stability.

SUMMARY:
The importance of physical activity and exercise-based interventions in neuro-orthopaedic rehabilitation is undisputed. Yet, patients and clinicians do not implement minimally required doses of physical activity in standard rehabilitation programs. This is partly due to intrinsic factors such as motivation, or due to physical condition that prevent any kind of exercise. In most cases, however, it is owed to limited time spent with therapists who would be able to supervise and apply the required doses to induce any potential exercise effects. Methods to semi-autonomously exercise with high motivation and continuous feedback would complement existing therapies and allow adherence to minimal dose recommendations.

For this study, a prototype of a new portable training solution for intensive walking exercise with built-in sensor-technology and a smartphone interface will be tested regarding its usability and its efficiency in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* In-patients with non-specified pathological background
* At trial centre for at least 2 weeks
* If less than 4 weeks, willingness to visit clinic for the remaining exercise sessions.
* Must be able to walk independently (no or minimal gait impairment)
* Deemed fit for walking group exercise and other exercise (medical expert opinion).
* Cleared for low-intensity endurance exercise by treating physicians and therapists (medical expert opinion).
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* Health condition does not allow free movements of body segments (e.g. un-consolidated upper limb fracture)
* Contraindications to low-intensity endurance training (e.g. congestive heart failure, unstable angina, peripheral arterial occlusive disease).
* Fresh wounds around waist and trunk.
* Orthopaedic condition that limits walking ability (e.g. newly operated total hip replacement).
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable double-barrier method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, combined with mechanical barriers (e.g. condoms or diaphragms) or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant (derived from medical history),
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Usability | 3-4 weeks
  Participants will be asked to rate the perceived usability based on the System Usability Scale (SUS). SUS assesses perceived effectiveness (can users successfully achieve their objectives), information quality (how much effort and resource is expended in achieving those objectives) and general satisfaction (was the experience satisfactory). The SUS hast 10 items that can be rated on a 5-point likert scale. The items will be scored as follows:
  1. For odd-numbered items, user response-1. For even-numbered items 5-user response. This scales all values from 0 to 4 (with four being the most positive response). Ref: Jeff Sauro, measuring usability
  2. Add up the converted responses for each user and multiply that total by 2.5 (to convert the range of possible values from 0 to 100 instead of from 0 to 40).
  3. single missing values are replaced with a neutral 3. Normative values will be used to grade the achieved median score (A through D, with D being least acceptable grade).

SECONDARY OUTCOMES:
Usability: Assists | 3-4 weeks
  Each participant will have a list of tasks to be completed per session. Amount of additional assistance following the introduction (after three supervised sessions), will be counted as outcome. E.g. additional verbal cues or practical assistance.
Usability: Completion rate efficiency [%/s] | 3-4 weeks
  Each participant will have a list of tasks to be completed per session. mean completion rate/mean task time = completion rate efficiency [%/s]; e.g. 80% completed all tasks within an average of 360 seconds.
  Task time: mean time taken before training was started [s].
Usability: Goal achievement efficiency [%/s] | 3-4 weeks
  Each participant will have a list of tasks to be completed per session. mean goal achievement/mean task time = Goal achievement efficiency [%/s]; e.g. 43% completed in 360 seconds Mean goal achievement: Mean extent to which the tasks were completed [%], e.g. 3 out of 7 tasks completed correctly = 43%.
Proof-of-Concept: Measurement of covered walking distance with the built-in sensors. | At first visit (t+0) and prior to first training 2-4 days after first vist (t+2)
  Standardised clinical assessment often employed as part of routine assessments will be used. The 10 Meter Walk Test (10MWT) is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Proof-of-Concept: Gait speed with the built-in sensors. | At first visit (t+0) and prior to first training 2-4 days after first vist (t+2)
  A second standardised clinical assessment often employed as part of routine assessments will be used. The 6 Minute Walk Test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance.
Proof-of-Concept: Increased intensity during walking (VCO2/VO2 relationship) | At first visit (t+0 days) and prior to first training 2-4 days after first vist (t+2 days)
  Cardiopulmonary response will be measured using a breath-by-breath cardiorespiratory monitoring system (MetaMax 3B, Cortex Biophysik, Leipzig, Germany) and a receiver board (HRMI, Sparkfun, Boulder, USA). During 10 meter walk test and a 6-minute walk test, oxygen uptake (VO2) and carbon dioxide output (VCO2) will be recorded and reported and VCO2/VO2 relationship.
Proof-of-Concept: Increased intensity during walking (heart rate) | At first visit (t+0 days) and prior to first training 2-4 days after first vist (t+2 days)
  During 10 meter walk test and a 6-minute walk test, heart rate (HR) will be recorded in both conditions (with and without belt). HR will be recorded over a rate belt (T31, Polar Electro, Kempele, Finland).

OTHER OUTCOMES:
Experience with walking exercises | At first visit (t+0 days).
  The amount of experience with walking exercise (qualitative, verbal description or as hours/week, if applicable),
General attitude towards technology based exercise: | At first visit (t+0 days).
  - attitude towards technology and the use of sensors (visual analogue scale, VAS, 0 to 100mm, where 0 stands for 'negative attitude' and 100 for 'positive attitude'),
Demographics: Age | At first visit (t+0 days).
  Age in years.
Demographics: Weight and height reported as BMI [kg/m^2] | At first visit (t+0 days).
  Weight [kg] and height [m] in BMI [kg/m^2]
Demographics: Profession | At first visit (t+0 days).
  Profession (qualitative description)
Attrition | 3 to 4 weeks after first visit.
  For attrition, the number of participants lost during the intervention was recorded. For adherence, participants' engagement with the intervention will be assessed.
Adherence | 3 to 4 weeks after first visit.
  Adherence will be calculated as the number of completed training sessions as a percentage of the maximal possible training sessions.
Exercise diary: | 3-4 weeks
  Training duration and intensity will be derived from the smartphone interface.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Behrendt, PhD, Principal Investigator — Reha Rheinfelden
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No